CLINICAL TRIAL: NCT03219775
Title: A Phase II Single Arm Clinical Trial of a Tailored ImmunoTherapy Approach With Nivolumab in Subjects With Metastatic or Advanced Transitional Cell Carcinoma
Brief Title: Tailored ImmunoTherapy Approach With Nivolumab in Subjects With Metastatic or Advanced Transitional Cell Carcinoma
Acronym: TITAN-TCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0416-ASG
Record Dates: First submitted 2017-07-04; First posted 2017-07-18 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Transitional Cell Carcinoma; Advanced Cancer; Metastatic Cancer
Keywords: tailored immuno therapy; Nivolumab; Ipilimumab; boost
MeSH Terms: conditions — Carcinoma, Transitional Cell; Neoplasm Metastasis | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab/Ipilimumab (Experimental): * Induction: Mono-Therapy with Nivolumab
  * If CR/PR: Nivolumab Maintenance Mono-Therapy
  * If SD/PD: Nivolumab/Ipilimumab "Boost 1+2"-Combination Therapy
  * If CR/PR: Nivolumab Maintenance Mono-Therapy
  * If SD/PD: Nivolumab/Ipilimumab "Boost 3+4"-Combination Therapy
  * If CR/PR/SD: Nivolumab Maintenance Mono-Therapy
  Interventions: Biological: Nivolumab/Ipilimumab

INTERVENTIONS:
Biological: Nivolumab/Ipilimumab — * Induction: Mono-Therapy with Nivolumab (240 mg i.V. / Q2W x 4)
  * If CR/PR: Nivolumab Maintenance Mono-Therapy (240 mg i.V. / Q2W)
  * If SD/PD: Nivolumab/Ipilimumab "Boost 1+2"-Combination Therapy (Nivo1 mg/kg i.V. and Ipi3 mg/kg i.V. / Q3W x 2)*
  * If CR/PR: Nivolumab Maintenance Mono-Therapy (240 mg i.V. / Q2W)
  * If SD/PD: Nivolumab/Ipilimumab "Boost 3+4"-Combination Therapy (Nivo 1 mg/kg i.V. and Ipi 3 mg/kg i.V. / Q3W x 2)
  * If CR/PR/SD: Nivolumab Maintenance Mono-Therapy (240 mg i.V. / Q2W)
    * since June 5, 2019, the treatment in all four "boost" cycles (1+2) and (3+4) is performed with nivolumab 1 mg/kg + ipilimumab 3 mg/kg (NIVO1/IPI3)
  Other Names: Opdivo/Yervoy

SUMMARY:
TITAN-TCC (0416-ASG) is a Phase 2, open-label study of nivolumab (BMS-936558) monotherapy with additional nivolumab/ipilimumab "boost" cycles in previously untreated* and platinum-based pretreated, 2nd and 3rd line, advanced or metastatic transitional cell carcinoma subjects. Nivolumab is a fully human PD-1 antibody which blocks the respective immune checkpoint in a ligand (PD-L1/PD-L2) independent manner.

[*Update from Jan-2020: First-line cohort was stopped and the inclusion of these patients was terminated]

DETAILED DESCRIPTION:
This is a Phase 2, single arm study of a tailored immunotherapy approach with nivolumab in adult (≥ 18 years) subjects with previously untreated (1st line)* or pretreated (2nd and 3rd line), surgically unresectable or metastatic TCC (further designated "advanced TCC"). The study targets to recruit 130 untreated (1st line) and 120 pretreated (2nd / 3rd line) patients, respectively. Tumor tissue obtained at least 2 years prior to screening must be available for a central pathology assessment. Subjects must have advanced (not amenable to curative surgery or radiation) or metastatic TCC, and must not have received more than two prior platinum-based chemotherapies for the treatment of advanced TCC.

[*Update from Jan-2020: First-line cohort was stopped and the inclusion of these patients was terminated. According protocol v.5.0 80 2nd/3rd-line patients need to be included]

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent

  * Subjects or legally acceptable representatives must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care.
  * Subjects or legally acceptable representatives must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study.
* Target Population

  * Histological evidence of metastatic or surgically unresectable transitional cell carcinoma of the bladder, urethra, ureter, or renal pelvis. Minor histologic variants of transitional cell carcinoma (e.g. squamous cell, comprising <50 % of the tumor overall) are acceptable.
  * Subjects must have advanced or surgically unresectable TCC (cT4b, any N or any T, N2-N3 or any M1) or having progressed during or after platinum-based first line therapy and up to 1 further treatment line (2nd and 3rd line cohort). Subjects, who have received neoadjuvant or adjuvant cisplatin based chemotherapy are eligible and considered first line provided that progression has occurred >12 months from last therapy [for chemoradiation and adjuvant treatment] or >12 months from last surgery [for neoadjuvant treatment]; in all other patients who received cisplatin based neoadjuvant and/or adjuvant chemotherapy and progression within 12 months this will be considered one line of therapy. [*Update January 2020:First-line cohort has been stopped since 31-Jan-2019 and wont be restarted]
  * KPS of at least 70% (See Appendix 1)
  * Measurable disease as per RECIST v1.1 (See Appendix 2)
  * Formalin-fixed paraffin embedded tumor tissue obtained within 2 years prior to screening must be available and received by the central pathology (tumor block is preferred, alternatively 15 unstained slides). Note that:

    1. Fine Needle Aspiration [FNA] and bone metastases samples (without soft tissue component) are not acceptable for submission).
    2. Tumor lesions used for newly acquired biopsies should not be target lesions, unless there are no other lesions.
* Age and Reproductive Status

  * Males and Females, ≥ 18 years of age
  * Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.
  * Women must not be breastfeeding
  * Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception for a period of 30 days (duration of ovulatory cycle) plus the time required for the investigational drug to undergo five half lives. The terminal half lives of nivolumab and ipilimumab are up to 25 days and 18 days, respectively. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug.
  * Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for a period of 90 days (duration of sperm turnover) plus the time required for the investigational drug to undergo five half lives. The terminal half lives of nivolumab and ipilimumab are up to 25 days and 18 days, respectively. Males who receive nivolumab combined with ipilimumab who are sexually active with WOCBP must continue contraception for 31 weeks (90 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug.

    * Comment: Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, WOCBP must still undergo pregnancy testing as described in this section.

Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy Investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly.

At a minimum, subjects must agree to the use of two methods of contraception, with one method being highly effective and the other method being either highly effective or less effective as listed below:

HIGHLY EFFECTIVE METHODS OF CONTRACEPTION

* Male condoms with spermicide
* Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants and intrauterine devices (IUDs) such as Mirena® by WOCBP subject or male subject's WOCBP partner. Female partners of male subjects participating in the study may use hormone based contraceptives as one of the acceptable methods of contraception since they will not be receiving study drug
* Nonhormonal IUDs, such as ParaGard®
* Tubal ligation
* Vasectomy
* Complete Abstinence*

  * *Complete abstinence is defined as complete avoidance of heterosexual intercourse and is an acceptable form of contraception for all study drugs. Subjects who choose complete abstinence are not required to use a second method of contraception, but female subjects must continue to have pregnancy tests. Acceptable alternate methods of highly effective contraception must be discussed in the event that the subject chooses to forego complete abstinence.

LESS EFFECTIVE METHODS OF CONTRACEPTION

* Diaphragm with spermicide
* Cervical cap with spermicide
* Vaginal sponge
* Male Condom without spermicide
* Progestin only pills by WOCBP subject or male subject's WOCBP partner
* Female Condom*.

  * * A male and female condom must not be used together

Exclusion Criteria:

* Target Disease Exceptions

  * Any history of or current CNS metastases. Baseline imaging of the brain by MRI (preferred) or CT scan is required within 28 days prior to registration in 2nd/3rd line patients only.
* Medical History and Concurrent Diseases

  * Prior systemic treatment with more than two different chemotherapy regimen (Sequential chemotherapy as a planned sequence to optimize response will count as 1 regimen)
  * Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti CTLA 4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
  * Any active or recent history of a known or suspected autoimmune disease or recent history of a syndrome that required systemic corticosteroids (> 10 mg daily prednisone equivalent) or immunosuppressive medications except for syndromes which would not be expected to recur in the absence of an external trigger. Subjects with vitiligo or type I diabetes mellitus or residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement are permitted to enroll.
  * Any condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to first dose of study drug. Inhaled steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
  * Prior malignancy active within the previous 3 years except for

    1. locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
    2. Patients in active surveillance for prostate cancer
  * Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS).
  * Any positive test for hepatitis B or hepatitis C virus indicating acute or chronic infection.
  * Known medical condition (eg, a condition associated with diarrhea or acute diverticulitis) that, in the investigator's opinion, would increase the risk associated with study participation or study drug administration or interfere with the interpretation of safety results.
  * Major surgery (eg, nephrectomy) less than 28 days prior to the first dose of study drug.
  * Anti-cancer therapy less than 28 days prior to the first dose of study drug or palliative, focal radiation therapy less than 14 days prior to the first dose of study drug.
  * Presence of any toxicities attributed to prior anti-cancer therapy other than neuropathy, alopecia and fatigue, that have not resolved to Grade 1 (NCI CTCAE v4) or baseline before administration of study drug.
* Physical and Laboratory Test Findings

  * Any of the following laboratory test findings:

    1. WBC < 2,000/mm^3
    2. Neutrophils < 1,500/mm^3
    3. Platelets < 100,000/mm^3
    4. AST or ALT > 3 x ULN (> 5 x ULN if liver metastases are present)
    5. Total Bilirubin > 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
    6. Serum creatinine > 1.5 x upper limit of normal (ULN) or creatinine clearance < 40 mL/min (measured or calculated by Cockroft-Gault formula):

       * Female CrCl = [(140 - age in years) x weight in kg x 0.85] / [72 x serum creatinine in mg/dL]
       * Male CrCl = [(140 - age in years) x weight in kg x 1.00] / [72 x serum creatinine in mg/dL]
* Allergies and Adverse Drug Reaction

  * History of severe hypersensitivity reaction to any monoclonal antibody or any constituent of the products.
* Other Exclusion Criteria

  * Prisoners or subjects who are involuntarily incarcerated
  * Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness
  * Participation in another clinical intervention trial 30 days prior to registration

Eligibility criteria for this study have been carefully considered to ensure the safety of the study subjects and that the results of the study can be used. It is imperative that subjects fully meet all eligibility criteria.

Subject Re-enrollment: This study permits the re-enrollment of a subject that has discontinued the study as a pre-treatment failure (ie, subject has not been registered / has not been treated). If re-enrolled, the subject must be re-consented.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2023-02-18 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | max. months
  The primary objective will be measured by the primary endpoint of ORR (based on investigator assessments) among all treated subjects, first line subjects and second line subjects. It is defined as the number of subjects with a best overall response of CR or PR divided by the number of all treated subjects, first line subjects or second line subjects. Best overall response is defined as the best response designation, as determined by investigator, recorded between the date of first dose and the date of objectively documented immunotherapy resistance per RECIST v1.1 or the date of subsequent therapy, whichever occurs first.

SECONDARY OUTCOMES:
Remission Rates (RR) | max. 68 months
  Remission Rates (RR) during TITAN treatment: CR/PR
Time to Immunotherapy Resistance (TIR) | max. 68 months
  Time to Immunotherapy Resistance (TIR) will be used as a surrogate parameter of progression free survival using a tailored Immunotherapy regimen with "boost" cycles upon initial progression.
Time to Response (TTR) | max. 68 months
  TTR is defined either as the time from first dosing date or initiation of nivolumab/ipilimumab "boost" cycles to the date of the first confirmed response thereafter, as assessed by the IRC. Hence, TTR may be recorded several times per patient.
Duration of Response (DOR) | max. 68 months
  DOR is defined as the time from first confirmed response (CR or PR) to the date of the documented progressive disease as determined using RECIST 1.1 criteria or death due to any cause, whichever occurs first. DOR may be recorded multiple times per patient.
Progression free survival (PFS) | max. 68 months
  PFS is defined as the time from first dosing date to the date of the first documented tumor progression based on investigator assessments (per RECIST 1.1), or death due to any cause. Clinical deterioration in the absence of unequivocal evidence of progression (per RECIST 1.1) is not considered progression for purposes of determining PFS.
Overall survival (OS) | max. 68 months
  OS is defined as the time from first dosing date to the date of death. A subject who has not died will be censored at last known date alive.
Safety - Incidence of adverse events, serious adverse events, deaths and laboratory abnormalities | max. 68 months
  Safety and tolerability objective will be measured by the incidence of adverse events, serious adverse events, deaths and laboratory abnormalities. Toxicities will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
EORTC QLQ-C30 | max. 68 months
  Questionaires
EQ-5D | max. 68 months
  Questionaires
EQ-5D VAS | max. 68 months
  Visual analogue scale

OTHER OUTCOMES:
Immune monitoring (Exploratory Endpoint) | max. 68 months
  Parameters will be analysed with regard to the prediction of response as well as immune related adverse events.
PD-L1 and PD-L2 | max. 68 months
  the expression of PD-L1 and PD-L2 in tumor tissues of mTCC patients will be correlated with efficacy parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Oliver Grimm, Prof. Dr., Principal Investigator — Jena University Hospital
Locations (27):
- Austria (5):
  - Univ. Klinik für Innere Medizin, Graz
  - Ordensklinikum Linz - KH Barmherzige Schwestern, Linz
  - Universitätsklinikum Salzburg, Salzburg
  - KH der Barmherzigen Brüder Wien, Vienna
  - Landesklinikum Wiener Neustadt, Wiener Neustadt
- Germany (22):
  - Universitätsklinikum Jena und Poliklinik für Urologie, Jena, Thuringia
  - Uniklinik der RWTH Aachen, Aachen
  - Vivantes Klinikum Neukölln, Berlin
  - Studienzentrum Bayenthal, Cologne
  - Uniklinik C.-G.-Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Helios Klinikum Erfurt, Erfurt
  - Universitätsklinikum Erlangen, Erlangen
  - Chirurgische Universitätsklinik Freiburg, Freiburg im Breisgau
  - Überörtliche Gemeinschaftspraxis für Urologie GbR, Fürth
  - Greifswald Universitätsklinikum, Greifswald
  - Universitätsklinikum Heidelberg Chirurgische Klinik Klinik für Urologie, Heidelberg
  - Marien Hospital, Herne
  - Urologie Herzberg, Herzberg am Harz
  - Universitätsklinikum Magdeburg, Magdeburg
  - UKGM Marburg, Marburg
  - Klinikum der Universität München - Großhadern, München
  - Universitätsklinikum Münster, Münster
  - Universtätsmedizin Rostock, Rostock
  - Universitätsklinikum Ulm, Ulm
  - Kliniken Nordoberpfalz AG, Klinikum Weiden, Weiden
  - Urologie Praxis am Wasserturm, Würselen

REFERENCES:
- [Derived] Grimm MO, Schostak M, Grun CB, Loidl W, Pichler M, Zimmermann U, Schmitz-Drager B, Steiner T, Roghmann F, Niegisch G, Bolenz C, Schmitz M, Baretton G, Leucht K, Schumacher U, Foller S, Zengerling F, Meran J; TITAN-TCC Study Group. Nivolumab + Ipilimumab as Immunotherapeutic Boost in Metastatic Urothelial Carcinoma: A Nonrandomized Clinical Trial. JAMA Oncol. 2024 Jun 1;10(6):755-764. doi: 10.1001/jamaoncol.2024.0938. PMID 38722641
- [Derived] Grimm MO, Grun CB, Niegisch G, Pichler M, Roghmann F, Schmitz-Drager B, Baretton G, Schmitz M, Bolenz C, Foller S, Leucht K, Schumacher U, Schostak M, Meran J, Loidl W, Zengerling F. Tailored immunotherapy approach with nivolumab with or without ipilimumab in patients with advanced transitional cell carcinoma after platinum-based chemotherapy (TITAN-TCC): a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2023 Apr;24(4):347-359. doi: 10.1016/S1470-2045(23)00053-0. Epub 2023 Feb 28. PMID 36868252
- [Derived] Grimm MO, Schmitz-Drager BJ, Zimmermann U, Grun CB, Baretton GB, Schmitz M, Foller S, Leucht K, Schostak M, Zengerling F, Schumacher U, Loidl W, Meran J. Tailored Immunotherapy Approach With Nivolumab in Advanced Transitional Cell Carcinoma. J Clin Oncol. 2022 Jul 1;40(19):2128-2137. doi: 10.1200/JCO.21.02631. Epub 2022 Mar 11. PMID 35275706